CLINICAL TRIAL: NCT01102374
Title: Vitamin D Supplementation and Acute Respiratory Infection in Older Long-Term Care Residents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH); The American Geriatrics Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 09-0899; IND 106541 (Other: FDA); K23AG040708 (NIH)
Record Dates: First submitted 2010-04-11; First posted 2010-04-13 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Respiratory Infection
Keywords: Vitamin D Deficiency; Respiratory Infection; Nursing Home Residents; Geriatrics; Immunosenescence; Prevention
MeSH Terms: conditions — Respiratory Tract Infections; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Dose Vitamin D (Experimental): 100,000 IU Vitamin D3 (cholecalciferol) monthly for 12 months. When added to usual care (0-1000 IU Vitamin D per day), averages 3,300-4,300 IU per day.
  Interventions: Drug: High Dose Vitamin D; Dietary Supplement: Usual Care
- Standard Dose Vitamin D (Active Comparator): 12,000 IU Vitamin D3 (cholecalciferol) or placebo monthly for 12 months. When added to usual care (0-1000 IU Vitamin D per day), averages 400-1,000 IU per day.
  Interventions: Drug: Standard Dose Vitamin D; Drug: Placebo; Dietary Supplement: Usual Care

INTERVENTIONS:
Drug: High Dose Vitamin D — Vitamin D3 100,000 IU monthly
  Arms: High Dose Vitamin D
Drug: Standard Dose Vitamin D — Vitamin D 12,000 IU monthly
  Arms: Standard Dose Vitamin D
Drug: Placebo — Placebo monthly
  Arms: Standard Dose Vitamin D
Dietary Supplement: Usual Care — Usual care of 0-1000 IU vitamin D daily. This is present in both study arms.

SUMMARY:
This study will test the role of high dose vitamin D supplementation in prevention of acute respiratory infection in older nursing home residents. The investigators hypothesize that residents on high dose vitamin D supplementation will have a lower incidence of acute respiratory infection that those on standard dose vitamin D supplementation.

DETAILED DESCRIPTION:
This study is a double-blinded, parallel group, randomized controlled phase II trial of oral high vs. standard dose vitamin D3 supplementation administered monthly for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 60+ years
* Resides in nursing home

Exclusion Criteria:

* Terminal illness (expected survival <6 months)
* Anticipated discharge within 12 months
* Unable to take whole or crushed tablets
* Active cancer, except squamous/basal cell carcinoma
* Severe malnutrition (body mass index <18 kg/m2)
* Current immunosuppressive medications (including corticosteroids)
* Renal failure (estimated glomerular filtration rate < 15 mL/min/1.73m2)
* Currently taking >1,000 IU/d vitamin D supplementation
* History (or strong family history) of kidney stones
* History of sarcoidosis or other granulomatous disorders associated with hypercalcemia
* Elevated baseline hypercalcemia (albumin-adjusted serum calcium >10.5 mg/dL)
* Baseline serum 25OHD level ≥ 100 nmol/L
* Inability to provide informed consent and no available healthcare legally authorized representative
* Inability of participant or legally authorized representative to speak/understand English

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adit A Ginde, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ginde AA, Blatchford P, Breese K, Zarrabi L, Linnebur SA, Wallace JI, Schwartz RS. High-Dose Monthly Vitamin D for Prevention of Acute Respiratory Infection in Older Long-Term Care Residents: A Randomized Clinical Trial. J Am Geriatr Soc. 2017 Mar;65(3):496-503. doi: 10.1111/jgs.14679. Epub 2016 Nov 16. PMID 27861708

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Started | 55 | 52
Completed | 39 | 33
Not Completed | 16 | 19
Not completed — Death | 9 | 13
Not completed — Lost to Follow-up | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D | Total
Number analyzed (Participants) | 55 | 52 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 80 (10) | 82 (10) | 81 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 29 | 62
  Male | 22 | 23 | 45
Region of Enrollment [Number; unit: participants]
  United States | 55 | 52 | 107
25-hydroxyvitamin D level [Mean (Standard Deviation); unit: ng/ml] | 23.0 (8.4) | 23.0 (9.9) | 23.0 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Acute Respiratory Infections (ARIs)
Description: ARIs defined as upper or lower respiratory infections
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 55 | 52
events | 32 | 48

2. Secondary Outcome: Severity of Acute Respiratory Infections
Description: ARIs resulting in emergency department visits or hospitalizations
Time Frame: 12 month
Measure: Number; unit: events
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 55 | 52
events | 3 | 6

3. Secondary Outcome: Time to First ARI
Time Frame: 12 months
Measure: Number; unit: Hazard Ratio
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 55 | 52
Hazard Ratio | 0.59 | 1.00

4. Secondary Outcome: Change in 25-hydroxyvitamin D (25OHD) Level
Time Frame: Baseline and 12 months
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 55 | 52
ng/mL | 8.18 (0.75) | 2.71 (0.80)

5. Secondary Outcome: Change in Parathyroid Hormone Level
Time Frame: Baseline and 12 months
Population: Issue relating to sample collection/processing precluded measurement of PTH level in the trial
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Falls
Time Frame: 12 months
Measure: Number; unit: Events
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 55 | 52
Events | 70 | 27

7. Secondary Outcome: Fractures
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 55 | 52
events | 5 | 8

8. Secondary Outcome: Number of Upper Respiratory Infections
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 55 | 52
events | 21 | 36

9. Secondary Outcome: Number of Lower Respiratory Infections
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 55 | 52
events | 11 | 12

10. Secondary Outcome: Number of Influenza-like Illnesses
Time Frame: 12 months
Population: collected together with lower respiratory infections (not as a separate category)
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Incident Kidney Stones
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 55 | 52
Participants | 0 | 0

12. Secondary Outcome: Incident Hypercalcemia
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 55 | 52
Participants | 0 | 0

13. Secondary Outcome: Death
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 55 | 52
Participants | 9 | 13

14. Secondary Outcome: Number of Urinary Tract Infections
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 55 | 52
events | 38 | 22

15. Secondary Outcome: Number of Other Infections
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Number analyzed (Participants) | 55 | 52
events | 33 | 43

ADVERSE EVENTS:
Arm/Group | High Dose Vitamin D | Standard Dose Vitamin D
Serious Adverse Events (participants affected / at risk) | 9/55 | 13/52
Other Adverse Events (participants affected / at risk) | 53/55 | 49/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Vitamin D (N=55) | Standard Dose Vitamin D (N=52)
Death (General disorders) | 9 (9) | 13 (13)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Vitamin D (N=55) | Standard Dose Vitamin D (N=52)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 7 | 4 — Adverse events were recorded at the organ system level using the MedDRA classification system
Cardiac disorders (Cardiac disorders) | 15 | 9 — Adverse events were recorded at the organ system level using the MedDRA classification system
Ear and labyrinth disorders (Ear and labyrinth disorders) | 6 | 1 — Adverse events were recorded at the organ system level using the MedDRA classification system
Endocrine disorders (Endocrine disorders) | 3 | 0 — Adverse events were recorded at the organ system level using the MedDRA classification system
Eye disorders (Eye disorders) | 5 | 7 — Adverse events were recorded at the organ system level using the MedDRA classification system
Gastrointestinal disorders (Gastrointestinal disorders) | 22 | 27 — Adverse events were recorded at the organ system level using the MedDRA classification system
General disorders (General disorders) | 39 | 28 — Adverse events were recorded at the organ system level using the MedDRA classification system
Hepatobiliary disorders (Hepatobiliary disorders) | 1 | 1 — Adverse events were recorded at the organ system level using the MedDRA classification system
Immune system disorders (Immune system disorders) | 9 | 7 — Adverse events were recorded at the organ system level using the MedDRA classification system
Infections and infestations (Infections and infestations) | 21 | 21 — Adverse events were recorded at the organ system level using the MedDRA classification system
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 29 | 30 — Adverse events were recorded at the organ system level using the MedDRA classification system
Investigations (Investigations) | 16 | 12 — Adverse events were recorded at the organ system level using the MedDRA classification system
Metabolic and nutrition disorders (Metabolism and nutrition disorders) | 18 | 15 — Adverse events were recorded at the organ system level using the MedDRA classification system
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 17 | 16 — Adverse events were recorded at the organ system level using the MedDRA classification system
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 — Adverse events were recorded at the organ system level using the MedDRA classification system
Nervous system disorders (Nervous system disorders) | 10 | 10 — Adverse events were recorded at the organ system level using the MedDRA classification system
Psychiatric disorders (Psychiatric disorders) | 30 | 19 — Adverse events were recorded at the organ system level using the MedDRA classification system
Renal and urinary disorders (Renal and urinary disorders) | 13 | 10 — Adverse events were recorded at the organ system level using the MedDRA classification system
Reproductive system disorders (Reproductive system and breast disorders) | 6 | 2 — Adverse events were recorded at the organ system level using the MedDRA classification system
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 24 | 30 — Adverse events were recorded at the organ system level using the MedDRA classification system
Skin and subcutaneous disorders (Skin and subcutaneous tissue disorders) | 23 | 22 — Adverse events were recorded at the organ system level using the MedDRA classification system
Social circumstances (Social circumstances) | 1 | 0 — Adverse events were recorded at the organ system level using the MedDRA classification system
Surgical and medical procedures (Surgical and medical procedures) | 14 | 6 — Adverse events were recorded at the organ system level using the MedDRA classification system

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No